CLINICAL TRIAL: NCT00977301
Title: The Effect of FOsamprenavir/Ritonavir on the Pharmacokinetics of a Single-dose of the Antipsychotic Agent olanZApine (FORZA)
Brief Title: Interaction Between Fosamprenavir/Ritonavir and a Single-dose Olanzapine (FORZA)
Acronym: FORZA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: D.M. Burger, PharmD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 08.04
Record Dates: First submitted 2009-08-17; First posted 2009-09-15 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections
Keywords: HIV infection; interaction; pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — fosamprenavir; Ritonavir; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fosamprenavir/ritonavir/olanzapine (Experimental): single dose of 15 mg olanzapine after 13 days of fosamprenavir/ritonavir 700mg/100mg BID
  Interventions: Drug: fosamprenavir/ritonavir; Drug: olanzapine
- single dose olanzapine (Active Comparator): Single dose of 10 mg olanzapine
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: fosamprenavir/ritonavir — 16 days 700mg/100mg RTV BID
  Arms: fosamprenavir/ritonavir/olanzapine
Drug: olanzapine — 15 mg olanzapine single dose
  Arms: fosamprenavir/ritonavir/olanzapine
Drug: olanzapine — 10 mg olanzapine single dose
  Arms: single dose olanzapine

SUMMARY:
The effect of fosamprenavir/ritonavir (steady state) on the pharmacokinetics of a single dose of olanzapine will be studied.

In this study, the investigators expect an inducible effect of fosamprenavir/ritonavir on the CYP1A2 and UGT metabolism of olanzapine.

DETAILED DESCRIPTION:
Psychosis and other mental illnesses are commonly described in patients infected with the human immunodeficiency virus (HIV). New-onset psychosis is estimated to occur in up to 15% of patients infected with HIV while 5 to 7% of patients with HIV-infection suffer from pre-existing mental illnesses including schizophrenia. Olanzapine could be an attractive antipsychotic in HIV/AIDS patients with schizophrenia.

Because olanzapine is a substrate for both UGT and CYP1A2, the pharmacokinetics of olanzapine might be influenced by low-dose ritonavir in combination with fosamprenavir. The current study is designed to test this hypothesis. Furthermore, in this study we evaluate the safety of such combination.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years at screening.
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electro-cardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to the first dose. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Pregnant female (as confirmed by an HCG test performed less than 4 weeks before the first dose) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the trial.
* Therapy with any drug (for two weeks preceding dosing), except for paracetamol.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, glaucoma, gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose.
* History of narrow-angle glaucoma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
olanzapine concentrations | pharmacokinetic curve after a single dose of olanzapine alone or added to steady state fosamprenavir/ritonavir

SECONDARY OUTCOMES:
adverse events | entire study

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- CRCN, Radboud Universtity Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Result] Jacobs BS, Colbers AP, Velthoven-Graafland K, Schouwenberg BJ, Burger DM. Effect of fosamprenavir/ritonavir on the pharmacokinetics of single-dose olanzapine in healthy volunteers. Int J Antimicrob Agents. 2014 Aug;44(2):173-7. doi: 10.1016/j.ijantimicag.2014.03.014. Epub 2014 May 23. PMID 24929949